CLINICAL TRIAL: NCT01699282
Title: Benefits of a Comprehensive Patient Education on Oral Anticoagulant Compared to Conventional Hospital Education.
Acronym: EDUCA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CHU-0121
Record Dates: First submitted 2012-07-13; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Cardiac Surgery
Keywords: oral anticoagulant; in the long term (> 12 months)
MeSH Terms: interventions — Educational Status

ARMS (2):
- Group thorough VKA (antivitamin K)education (Experimental)
  Interventions: Behavioral: VKA (antivitamin K) education
- control group (Active Comparator)
  Interventions: Behavioral: conventional hospital education

INTERVENTIONS:
Behavioral: VKA (antivitamin K) education — Evaluate benefits of a comprehensive patient education on oral anticoagulant compared to conventional hospital education
  Arms: Group thorough VKA (antivitamin K)education
Behavioral: conventional hospital education — Group thorough VKA education V.S. control group (conventional hospital education)
  Arms: control group

SUMMARY:
To meet the wishes of the Ministry of Health, the division of Cardiology University Hospital of Clermont Ferrand, combining the cardiology and cardiac surgery department, has developed since January 2009, a therapeutic education to use oral anticoagulants, in collaboration with the functional rehabilitation center Durtol. All patients under VKA, are formed by nurses. The purpose of this local study, in cardiac surgery department, is to evaluate the therapeutic impact of two methods of comprehensive education, one conventional and performed by nurses service, less elaborate, relying solely on the book Information from The National Security Agency of Medicines and Health Products, the other based on more detailed documents created by a multidisciplinary group. Various studies show that the effect of therapeutic education is observed only during the first six months and then disappears.

This study is the first French study evaluating the impact of a comprehensive education to oral anticoagulation according to the latest recommendations of the National Security Agency of Medicines and Health Products and the French National Health Authority.

DETAILED DESCRIPTION:
To meet the wishes of the Ministry of Health, the division of Cardiology University Hospital of Clermont Ferrand, combining the cardiology and cardiac surgery department, has developed since January 2009, a therapeutic education to use oral anticoagulants, in collaboration with the functional rehabilitation center Durtol. All patients under VKA, are formed by nurses. The purpose of this local study, in cardiac surgery department, is to evaluate the therapeutic impact of two methods of comprehensive education, one conventional and performed by nurses service, less elaborate, relying solely on the book Information from The National Security Agency of Medicines and Health Products, the other based on more detailed documents created by a multidisciplinary group. Various studies show that the effect of therapeutic education is observed only during the first six months and then disappears.

This study is the first French study evaluating the impact of a comprehensive education to oral anticoagulation according to the latest recommendations of the National Security Agency of Medicines and Health Products and the French National Health Authority.

ELIGIBILITY:
Inclusion Criteria:

* Adults, male or female, over 18 years
* After cardiac surgery
* Requiring an oral anticoagulant in the long term (> 12 months)
* Accepting the principle of extended follow-up
* Voluntary Consent, written and signed by patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
knowledge test on anticoagulant treatment | after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kasra Azarnoush, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France